CLINICAL TRIAL: NCT02247843
Title: Clinical Research Study of Autologous Stem Cell Transplantation for Sickle Cell Disease (SCD) Using Peripheral Blood CD34+ Cells Modified With the Lenti/G-βAS3-FB Lentiviral Vector
Brief Title: Stem Cell Gene Therapy for Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Donald B. Kohn, M.D. (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Donald B. Kohn, M.D., Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lenti/βAS3-FB
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease (SCD); Gene Therapy; Lentiviral Vector; Beta Globin
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- βAS3-FB vector transduced peripheral blood CD34+ cells (Experimental): This is a single arm study without randomization. All subjects will receive the intervention of BetaAS3 lentiviral vector-modified autologous peripheral blood stem cell transplant.
  Interventions: Biological: βAS3-FB vector transduced peripheral blood CD34+ cells

INTERVENTIONS:
Biological: βAS3-FB vector transduced peripheral blood CD34+ cells — CD34+ from the peripheral blood of patients with sickle cell disease (SCD) are transduced ex-vivo with the Lenti/βAS3-FB lentiviral vector. The transduced cells are then infused into the patient.
  Other Names: Lenti/βAS3-FB

SUMMARY:
This Phase I clinical trial will assess the safety and initial evidence for efficacy of an autologous transplant of lentiviral vector modified peripheral blood for adults with severe sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) affects ~90,000 people in the U.S. who suffer significant neurological, lung, and kidney damage, as well as severe chronic pain episodes that adversely impact on quality of life. While current medical therapies for SCD can reduce short-term morbidity, the inevitable progressive deterioration in organ function results in a significant decrease in quality of health with early mortality. Allogeneic hematopoietic stem cell transplant (HSCT) can benefit patients with SCD, by providing a source for life-long production of normal red blood cells. However, allogeneic HSCT is limited by the availability of well-matched donors and immunological complications, especially for the more than 80% of patients who lack an HLA-identical sibling donor. Autologous HSCT using a patient's own peripheral blood stem cells that have been corrected by transfer of a modified human beta-globin gene that inhibits polymerization of the HbS (stem cell gene therapy) may provide a better therapeutic alternative, as it would avoid the immunologic complications and donor limitations of allogeneic HSCT.

Up to 6 subjects with SCD meeting eligibility criteria for disease severity and adequacy of organ function will be enrolled.

Following informed consent, enrolled subjects will be screened to confirm full eligibility for participation. A chronic red blood cell transfusions regimen will be given prior to stem cell collection and transplant. Subjects will undergo peripheral blood stem cell collection using plerixafor mobilization and apheresis. A portion of their stem cells will be cryopreserved as "back-up," with the remaining portion used to prepare the gene-modified Final Cellular Product: autologous peripheral blood CD34+ cells transduced ex vivo by the Lenti/G-βAS3-FB lentiviral vector to express an anti-sickling (βAS3) gene. The subject will receive marrow cytoreduction with busulfan prior to infusion of the gene-modified cells. The follow-up period will include an initial 2 years of active follow-up, where the subjects will be seen at intervals of no more than 3 months, followed by offer for enrollment into a long-term follow-up study during years 3-15.

The primary objectives of the Phase I study are to assess safety and feasibility, with secondary objectives to assess efficacy (engraftment, βAS3-globin gene expression, and effects on red blood cells function and clinical hematologic and disease parameters).

ELIGIBILITY:
PARTICIPANT INCLUSION CRITERIA

* Age ≥18 by time of enrollment
* Diagnosis of SCD documented by genetic analysis (S/S, S/β-thalassemia-zero)
* Must not have medically eligible and available HLA-identical sibling donor or 10/10 allele-matched unrelated donor (within a year prior to harvest) (or refuses to have an allogeneic HSCT)
* Inadequate clinical response to hydroxyurea (HU), defined as any one of the following outcomes, while on HU for at least 3 months:

  * 2 or more acute sickle pain crises requiring hospitalization
  * no rise in Hb >1.5 gm/dl from pre-HU baseline or requires transfusion to maintain Hb > 6.0 gm/dL
  * Has an episode of acute chest syndrome defined as development of a new pulmonary alveolar consolidation involving at least one complete lung segment associated with acute symptoms including: fever >38.5, chest pain, tachypnea, intercostal retractions, nasal flaring, use of accessory muscles of respiration, wheezing, rales, or cough not attributable to asthma or bronchiolitis) in the preceding two year period prior to enrollment. The acute chest syndrome event occurred despite adequate supportive care measures.
  * Or medical decision for other therapy (e.g. chronic transfusion program), or subject refusal to take HU.
* The patient must be off HU for at least 30 days (+/- 5 days) before PBSC collection.
* Must have one or more of the following clinical complications demonstrating disease severity:

  * Clinically-significant neurologic event: stroke or any central nervous system deficit lasting >24 hours.
  * Abnormal head CT or brain MRI demonstrating previous stroke
  * Administration of regular RBC transfusions for equal or longer than 1 year to prevent vaso- occlusive crises or other sickle cell disease complications or to maintain Hb >6.
  * Pulmonary arterial hypertension with tricuspid regurgitant jet velocity > 2.5 m/sec within 1 year prior to enrollment
  * At least one episode of acute chest syndrome that required hospitalization, within the 2 years prior to enrollment
  * At least 2 acute sickle pain crises requiring hospitalization within the 2 years prior to enrollment
  * Severe osteonecrosis
  * History of acute dactylitis during childhood
  * Recurrent priapism (2 or more episodes)
* Karnofsky performance score ≥60%

PARTICIPANT EXCLUSION CRITERIA

* Patient has a medically eligible and available HLA-identical sibling donor or 10/10 allele-matched unrelated donor (unless they refuse to have an allogeneic HSCT).
* Cardiac evaluation: left ventricular ejection fraction (LVEF) < 40% or LV shortening fraction < 26% by cardiac echocardiogram or by MUGA scan or clinically significant ECG abnormalities.
* Poorly controlled hypertension as determined by BP with systolic >135 or diastolic >95 mmHg despite treatment.
* Pulmonary evaluation: baseline oxygen saturation of <85% or DLCO< 40% (corrected for Hb)
* Renal evaluation: serum creatinine >1.5x upper limit of normal for age or GFR<60 mL/min/1.73 m2 within 90 days prior to PBSC collection.
* Hepatic evaluation: serum conjugated (direct) bilirubin > 2x upper limit of normal for age as per local laboratory or ALT and AST > 5 times upper limit of normal as per local laboratory within 90 days prior to PBSC collection.
* Hematologic evaluation: Leukopenia (WBC< 3x103/uL) or neutropenia (ANC < 1.0x103/uL) or thrombocytopenia (platelet count < 100x103/uL) within 90 days prior to PBSC collection.
* PT/INR or PTT >1.5x upper limit of normal or other clinically significant bleeding disorder to
* Liver Iron >10mg/g by T2* MRI (within 1 year prior to PBSC collection).
* Seropositivity for HIV (Human Immunodeficiency Virus), HCV (Hepatitis C Virus), HTLV-1 (Human T-Lymphotropic Virus), or active Hepatitis B Virus, or active infection by CMV or parvovirus B19, based on positive blood PCR.
* Pregnancy
* Patient must not have any known cancer or other malignant disease or active infection by CT or MRI of head, chest or ultrasound of abdomen
* Abnormal karyotype by cytogenetic or other appropriate tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety | up to 24 months
  1. Clinical toxicity: Absence of grade 3-4 SAEs
  2. Absence of replication-competent lentivirus (RCL):
  3. Absence of monoclonal expansion or leukoproliferative disorder from vector insertional effects: To monitor for monoclonal expansion or leukoproliferative complications, LAM-PCR will be performed.
  4. Event-free survival. Event-free survival will be determined for each subject over the 24 months after gene therapy. An event is defined as death or performance of an allogeneic HSCT.
  5. Absence of humoral immune response to novel epitopes of βAS3-globin protein

CONTACTS AND LOCATIONS:
Overall Officials: Donald Kohn, MD, Study Chair — University of California, Los Angeles; Gary Schiller, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero Z, Urbinati F, Geiger S, Cooper AR, Wherley J, Kaufman ML, Hollis RP, de Assin RR, Senadheera S, Sahagian A, Jin X, Gellis A, Wang X, Gjertson D, Deoliveira S, Kempert P, Shupien S, Abdel-Azim H, Walters MC, Meiselman HJ, Wenby RB, Gruber T, Marder V, Coates TD, Kohn DB. beta-globin gene transfer to human bone marrow for sickle cell disease. J Clin Invest. 2013 Jul 1;123(8):3317-30. doi: 10.1172/JCI67930. Online ahead of print. PMID 23863630